CLINICAL TRIAL: NCT05779254
Title: Analysis of Mechanism on the Efficacy of Oral Antibiotic Prophylaxis in Elective Colon and Rectal Surgery With Primary Anastomosis
Brief Title: SURGIcal COmplication and MIcrobiome ChangeS in Colorectal Surgery
Acronym: Surgi-Comics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uzsoki Hospital (Other)
Collaborators: University of Debrecen (Other); Csolnoky Ferenc Hospital (Unknown)
Responsible Party: Principal Investigator, Dr. Papp Géza, Principal Investigator, Uzsoki Hospital
Other Study IDs: Surgi-Comics_01
Record Dates: First submitted 2023-02-12; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Anastomotic Leak; Microbial Colonization
Keywords: Colorectal surgery; Anastomotic leak; Surgical site infection; Microbiome; Oral antibiotic prophylaxis
MeSH Terms: conditions — Anastomotic Leak; Communicable Diseases; Surgical Wound Infection | interventions — Neomycin; Metronidazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Anastomotic ring full thickness colonic wall
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oral Antibiotic Prophylaxis +: At the Uzsoki Hospital and the Department of Surgery at the University of Debrecen, patients receive preoperative neomycin- metronidazole oral antibiotic prophylaxis in addition to mechanical bowel preparation.
  Interventions: Drug: Neomycin Sulfate
- Oral Antibiotic Prophylaxis -: Patients admitted to the Csolnoky Ferenc Hospital in Veszprém will receive preoperative mechanical bowel preparation and no oral antibiotic prophylaxis.

INTERVENTIONS:
Drug: Neomycin Sulfate — Postoperative day-1 Oral Antibiotic Prophylaxis + patients get po. 3x1000mg Neomycin sulfate and 3x500 mg Metronidazole
  Other Names: Metronidazole
  Groups: Oral Antibiotic Prophylaxis +

SUMMARY:
The microbiome, the collection of microorganisms that live in our gut, plays an important role in maintaining our health, proper nutrient absorption, nutrient turnover and immunity. After birth, a symbiotic relationship develops with the strains of bacteria that colonise our gut, and the presence and proportion of bacteria is individualised and highly variable.

A healthy bacterial flora is essential for the cells of the intestinal mucosa. Glycoproteins in the cell surface mucus coat are important nutrients for bacteria, while some bacterial strains supply mucosal cells with nutrient molecules (e.g. short-chain fatty acids) that are their essential energy source.

An abnormal change in the proportion of bacterial strains that make up the microbiome, dysbacteriosis, in which pathogenic bacteria proliferate at the expense of members of the normal flora, can cause a number of pathologies. Nutrient supply to the cells of the mucosa is reduced, making them more vulnerable and leading to various pathological conditions.

The microbiome and the essential nutrients they produce have also been found to play an important role in wound healing. A decrease in the diversity of the microbiome, an increase in the relative number of pathogenic bacteria and a decrease in the proportion of 'beneficial' bacteria increases the risk of surgical complications of infection and suture failure.

DETAILED DESCRIPTION:
A number of risk factors have been identified that increase or decrease the risk of anastomotic leak. The risk of anastomotic failure is increased by anastomosis (lower third) close to the anus, tumour size greater than 5cm in colorectal carcinoma, surgical complications, smoking, diabetes, male gender, overweight, malnutrition (protein deficiency), heart disease requiring anticoagulation, time to surgery, American Society of Anaesthesiologist score, neoadjuvant treatment, corticosteroid use. The risk of suture failure is reduced by mechanical lining, intravenous and oral non-absorbable antibiotics. The microbiome also appears to have an impact on suture failure: lower diversity of bacteria in intraoperative specimens and an increase in the number of mucin-degrading Bacteroidaceae or Lachnospiraceae strains may be associated with higher anastomotic failure.

ELIGIBILITY:
Inclusion Criteria:

* Circular stapled anastomosis
* Planned surgery with colo-colic anastomosis
* No passage disorder, as it is confirmed at the first medical examination
* Not allergic to antibiotics
* Can receive a bowel preparation
* No proximal excluded intestine, i.e., the bowel preparation may be successful (ileostomy)

Exclusion Criteria:

* treated with antibiotics within 2 weeks before randomisation
* allergic to any of the medicines used
* under 18 years of age
* have suffered from abdominal sepsis within 6 months prior to recruitment
* pregnancy or breastfeeding
* been treated with steroids
* any form of chronic immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing planned colorectal surgery, whether open or laparoscopic, with circular suture anastomosis training are eligible for the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Microbiome | postoperative 30 days
  Is there evidence of a correlation between septic complications and the microbiome?

SECONDARY OUTCOMES:
Affecting factors on microbiome | postoperative 30 days
  Is it a relevant factor influencing the microbiome: comorbidities, previous operations, oral antibiotic prophylaxis, systemic intravenous prophylaxis?

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bay, Prof., Study Director — University of Debrecen
Locations (3):
- Hungary (3):
  - Uzsoki Hospital, Budapest
  - University of Debrecen, Debrecen
  - Csolnoky Ferenc Kórház, Veszprém

REFERENCES:
- [Background] Hajjar R, Santos MM, Dagbert F, Richard CS. Current evidence on the relation between gut microbiota and intestinal anastomotic leak in colorectal surgery. Am J Surg. 2019 Nov;218(5):1000-1007. doi: 10.1016/j.amjsurg.2019.07.001. Epub 2019 Jul 11. PMID 31320106
- [Background] van Praagh JB, de Goffau MC, Bakker IS, van Goor H, Harmsen HJM, Olinga P, Havenga K. Mucus Microbiome of Anastomotic Tissue During Surgery Has Predictive Value for Colorectal Anastomotic Leakage. Ann Surg. 2019 May;269(5):911-916. doi: 10.1097/SLA.0000000000002651. PMID 29303807
- [Background] Gaines S, Shao C, Hyman N, Alverdy JC. Gut microbiome influences on anastomotic leak and recurrence rates following colorectal cancer surgery. Br J Surg. 2018 Jan;105(2):e131-e141. doi: 10.1002/bjs.10760. PMID 29341151
- [Background] Nagata N, Tohya M, Fukuda S, Suda W, Nishijima S, Takeuchi F, Ohsugi M, Tsujimoto T, Nakamura T, Shimomura A, Yanagisawa N, Hisada Y, Watanabe K, Imbe K, Akiyama J, Mizokami M, Miyoshi-Akiyama T, Uemura N, Hattori M. Effects of bowel preparation on the human gut microbiome and metabolome. Sci Rep. 2019 Mar 11;9(1):4042. doi: 10.1038/s41598-019-40182-9. PMID 30858400
- [Background] Papp G, Saftics G, Szabo BE, Baracs J, Vereczkei A, Kollar D, Olah A, Meszaros P, Duboczki Z, Bursics A. Systemic versus Oral and Systemic Antibiotic Prophylaxis (SOAP) study in colorectal surgery: prospective randomized multicentre trial. Br J Surg. 2021 Apr 5;108(3):271-276. doi: 10.1093/bjs/znaa131. PMID 33793743
- [Background] Williamson AJ, Alverdy JC. Influence of the Microbiome on Anastomotic Leak. Clin Colon Rectal Surg. 2021 Nov 23;34(6):439-446. doi: 10.1055/s-0041-1735276. eCollection 2021 Nov. PMID 34853567
- [Background] Di Segni A, Braun T, BenShoshan M, Farage Barhom S, Glick Saar E, Cesarkas K, Squires JE, Keller N, Haberman Y. Guided Protocol for Fecal Microbial Characterization by 16S rRNA-Amplicon Sequencing. J Vis Exp. 2018 Mar 19;(133):56845. doi: 10.3791/56845. PMID 29608151
- [Background] Reuvers JRD, Budding AE, van Egmond M, Stockmann HBAC, Twisk JWR, Kazemier G, Abis GSA, Oosterling SJ; SELECT trial group. Gut Proteobacteria levels and colorectal surgical infections: SELECT trial. Br J Surg. 2023 Jan 10;110(2):129-132. doi: 10.1093/bjs/znac288. No abstract available. PMID 35998096